CLINICAL TRIAL: NCT03474991
Title: A Randomised Placebo-controlled Multi-centre Effectiveness Trial of Adjunct Betamethasone Therapy in Hospitalised Children With Community Acquired Pneumonia (CAP)
Brief Title: KIDS-STEP_Betamethasone Therapy in Hospitalised Children With CAP
Acronym: KIDS-STEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Julia Bielicki (Other)
Collaborators: Swiss National Fund for Scientific Research (Other); University Hospital, Basel, Switzerland (Other); SwissPedNet (Unknown)
Responsible Party: Sponsor-Investigator, Julia Bielicki, Sponsor-representative of University of Basel Children's Hospital (UKBB), University Children's Hospital Basel
Organization: University Children's Hospital Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-00563; me15CC7
Record Dates: First submitted 2018-03-16; First posted 2018-03-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: KIDS-STEP is a phase III strategic investigator-initiated, randomised, placebo-controlled, fully blinded multicentre superiority trial with two parallel groups
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Celestamine® N 0.5 (Active Comparator): oral betamethasone solution, once daily for two consecutive days at 0.1-0.2 mg/kg
  Interventions: Drug: Celestamine®
- Placebo (Placebo Comparator): oral placebo matched to the product described above
  Interventions: Drug: Celestamine®

INTERVENTIONS:
Drug: Celestamine® — Children in KIDS-STEP will be receiving either oral betamethasone (Celestamine®) or oral placebo dosed once daily for two consecutive days. Celestamine® N 0.5 liquidum is a betamethasone solution and will be used in the active comparator arm. Study medication will be administered orally once a day on two consecutive days. A standard dose of 0.1-0.2 mg/kg will be used. All doses used in KIDS-STEP fall into the range of recommended doses according to the Summary of Medical Product Characteristics.

SUMMARY:
The purpose of this study is to concurrently evaluate whether adjunct treatment with corticosteroids in children hospitalized with CAP is more effective in terms of the proportion of children reaching clinical stability and whether such adjunct treatment is no worse in terms of CAP relapse.

DETAILED DESCRIPTION:
The incidence of community-acquired pneumonia (CAP) in young children remains high (20- 30/1000 child-years) even in high-income settings with routine pneumococcal vaccination, and is associated with a high rate of hospitalisation (around 10/1000 child-years). In low-and middle-income settings, pneumonia is the leading infectious cause of death in children less than 5 years of age. In high-income settings, working mothers of children hospitalised with CAP have been reported to loose on average 4.2 workdays compared with 1.7 workdays for children with CAP managed in primary care. In addition to this economic burden, there is a substantial impact on quality of life for the affected child and the family. Children who are admitted with CAP experience on average 13 nonroutine days with slightly shorter periods of decreased appetite (8.5 days), disordered sleep (4.5 days) and absence from routine out-of-home childcare (7.5 days). Any intervention that ensures rapid clinical stabilization allowing for early hospital discharge without negative impacts on the overall recovery in children hospitalised with CAP would therefore carry substantial socioeconomic benefits.

Only few small trials have addressed the potential impact of oral steroid treatment in CAP during childhood. Nagy et al reported a significant reduction in fever duration and length of stay in children with severe CAP receiving methylprednisolone for 5 days compared with children receiving placebo in a randomised trial with 59 participants. A randomised trial comparing adjunct dexamethasone or methylprednisolone against standard of care (no placebo) planning to enroll 40 participants was being set up but has been withdrawn prior to recruitment (NCT01631916). A placebo-controlled randomised trial of adjunct corticosteroids in CAP complicated by pleural effusion and/or empyema with 56 participants has been completed (NCT01261546), but has not yet reported on its findings. An observational analysis using propensity scores found that adjunct corticosteroids were associated with a shorter hospital stay only in children also receiving beta-agonist therapy, concluding that any benefit might only be seen in children with acute wheezing. All in all, there is a lack of pragmatic randomized controlled trials ( RCT) with sufficient power and high external validity to provide a definitive answer to the question of the effect of adjunct steroids in children hospitalised with CAP.

Infection-related unwanted effects of adjunct steroids are potentially relevant in the context of childhood CAP. A higher proportion of children hospitalised with CAP reaching early clinical stability would only be desirable if this were shown not to be offset by a higher rate of clinically relevant CAP recurrence. A rebound phenomenon after corticosteroid discontinuation has been postulated to explain a higher rate of infection recurrence (19% compared with 9% in placebo group) among adults. Data from a recent individual patient data metaanalysis, however, indicate that an increased risk of CAP recurrence may be rather associated with longer duration of adjunct steroids in adults with CAP. To our knowledge, the question about the effect of adjunct steroid treatment in childhood CAP in relation to a postulated rebound phenomenon measured clinically as CAP recurrence has not been formally addressed in a trial. CAP-specific readmission rates for children are low at around 5%. In bronchiolitis, another acute lower respiratory tract infection for which oral corticosteroid treatment has been investigated, an increased risk of hospital revisits associated with steroid treatment could not be identified in a Cochrane metaanalysis.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 5 kg and 45 kg
* Admission to hospital (i.e. assignment of an inpatient case number)
* Clinical diagnosis of CAP (according to predefined criteria)
* Parent and/or child (as age-appropriate) willing to accept all possible randomised allocations and to be contacted by telephone weekly up to and including at 4 weeks after randomisation
* Informed consent form for trial participation signed by parent

Exclusion Criteria:

* Presence of local chest complications
* Chronic underlying disease associated with an increased risk of very severe CAP or CAP of unusual aetiology
* Bilateral wheezing without focal chest signs AND clinical indication for primary administration of steroids (most likely to represent respiratory tract infection affecting the medium airways, i.e. not pneumonia)
* Admission to hospital with a primary clinical diagnosis of bronchiolitis
* Inability to tolerate oral medication
* Documented allergy or any other known contraindication to any trial medication
* Subacute or chronic conditions requiring higher betamethasone equivalent or known primary or secondary adrenal insufficiency
* Known diabetes mellitus (type 1)
* Hospitalisation within the last two weeks preceding current admission with the possibility that pneumonia could be hospital-acquired or healthcare-associated
* Completion of a course of systemic corticosteroids within 2 weeks from enrolment for courses of >5 days
* Transfer for any reason to a non-participating hospital directly from the paediatric emergency department
* Parent are unlikely to be able to reliably participate in telephone follow-up because of significant language barriers
* Participation in another study with investigational drug within the 30 days preceding and during the present study
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, and other dependent persons.

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 510 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
time to clinical stability | from randomization up to 2 days
  The time to clinical stability after randomization in the active treated group (oral betamethasone for up to 2 days) as compared to the control group (placebo) will be one primary outcome.
CAP-related re-admission measured by number of childs re-admitted to hospital due to CAP | from randomization until day 28
  (ii) The proportion of children with CAP-related readmission within 28 days after randomization comparing oral betamethasone and placebo will be the co-primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes van der Anker, Prof MD, Principal Investigator — University of Basel Children's Hospital (UKBB)
Locations (13):
- Germany (4):
  - Universitätsklinikum der Ruhr-Universität Bochum, Klinik für Kinder- und Jugendmedizin, Bochum
  - Universitätsklinikum Düsseldorf, Klinik für Allgemeine Pädiatrie, Düsseldorf
  - Universitätsklinikum Freiburg, Zentrum für Kinder und Jugendmedizin Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Tübingen, Klinik für Kinder- und Jugendmedizin, Tübingen
- Switzerland (9):
  - Kantonsspital Aarau, Klinik für Kinder u. Jugendliche, Aarau
  - University of Basel Children's Hospital (UKBB), Basel
  - Inselspital Bern, Bern
  - Geneva University Hospital, Department of Pediatrics, Geneva
  - Centre hospitalier universitaire vaudois, Lausanne
  - Luzerner Kantonsspital, Kinderspital, Lucerne
  - Ostschweizer Kinderspital, Sankt Gallen
  - Kantonsspital- Freiburger Spital (HFR), Villars-sur-Glâne
  - University-Childrens Hospital Zürich, Zurich

REFERENCES:
- [Derived] Kohns Vasconcelos M, Meyer Sauteur PM, Keitel K, Santoro R, Heininger U, van den Anker J, Bielicki JA. Strikingly Decreased Community-acquired Pneumonia Admissions in Children Despite Open Schools and Day-care Facilities in Switzerland. Pediatr Infect Dis J. 2021 Apr 1;40(4):e171-e172. doi: 10.1097/INF.0000000000003026. No abstract available. PMID 33399433
- [Derived] Kohns Vasconcelos M, Meyer Sauteur PM, Santoro R, Coslovsky M, Lura M, Keitel K, Wachinger T, Beglinger S, Heininger U, van den Anker J, Bielicki JA. Randomised placebo-controlled multicentre effectiveness trial of adjunct betamethasone therapy in hospitalised children with community-acquired pneumonia: a trial protocol for the KIDS-STEP trial. BMJ Open. 2020 Dec 29;10(12):e041937. doi: 10.1136/bmjopen-2020-041937. PMID 33376176